CLINICAL TRIAL: NCT04433468
Title: Study on the Protective Effect of RIPC in Patients Undergoing Cardiac Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020RIPC
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Cardiac Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIPC (Active Comparator)
  Interventions: Device: RIPC
- Control (No Intervention)

INTERVENTIONS:
Device: RIPC — The tourniquet attached to the upper limb was inflated and blocked for 5 minutes, then deflated for 5 minutes to restore blood flow and induce ischemic preconditioning.
  Arms: RIPC

SUMMARY:
To observe the effect of RIPC on the function of vital organs after cardiac surgery, and to explore its possible mechanism.

ELIGIBILITY:
Inclusion Criteria:

* patients with aortic valve, mitral valve, tricuspid valve, ascending aortic disease and coronary atherosclerosis who were admitted to hospital for elective valve repair, replacement, artificial vascular replacement or coronary artery bypass grafting.
* age 18-80 years old.
* No restriction on gender.
* ASA grade II~III.
* NYHAII~III level.
* the patient or his family member has signed the informed consent form for the clinical trial

Exclusion Criteria:

* those who are disabled in the selected test.
* less than 5 years of education.
* The preoperative left ventricular ejection fraction ((LVEF)) was less than 40%.
* Myocardial infarction occurred in nearly one month.
* malignant tumor, hematological disease, severe liver and kidney dysfunction, recent severe infection, etc.
* History of nervous system, immune system and mental illness.
* recent operation history of heart, brain, lung, liver, kidney and other important organs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
The incidence of acute renal injury after operation | within 7 days after operation
  According to the (KDIGO) guidelines for improving the prognosis of renal disease
The incidence of postoperative delirium | within 7 days after operation
  CAM score greater than 22

CONTACTS AND LOCATIONS:
Locations (1):
- 180 Fenglin Road, Shanghai, China

IPD SHARING:
Plan to Share IPD: No